CLINICAL TRIAL: NCT03006887
Title: An Open-Label Phase 1b Trial of Lenvatinib Plus Pembrolizumab in Subjects With Selected Solid Tumors
Brief Title: Phase 1b Trial of Lenvatinib Plus Pembrolizumab in Participants With Selected Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-115; KEYNOTE 523 (Other: Merck)
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumors
Keywords: solid tumors; non-small cell lung cancer; predominantly clear cell renal cell carcinoma; endometrial carcinoma; urothelial carcinoma; squamous cell carcinoma of the head and neck; non-uveal melanoma; E7080; lenvatinib; pembrolizumab; Japan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Endometrial Neoplasms; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- lenvatinib 20 mg plus pembrolizumab 200 mg (Experimental): Participants with selected tumors will receive oral lenvatinib at a starting dose of 20 milligrams (mg) once daily in combination with intravenous pembrolizumab 200 mg every 3 weeks (Q3W) on a 21-day treatment cycle until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study.
  Interventions: Drug: lenvatinib; Drug: pembrolizumab

INTERVENTIONS:
Drug: lenvatinib — lenvatinib capsules
Drug: pembrolizumab — pembrolizumab intravenous infusion

SUMMARY:
This is an open-label Phase 1b study designed to confirm the tolerability and safety of lenvatinib in combination with pembrolizumab in participants with selected solid tumors (non-small cell lung cancer, predominantly clear cell renal cell carcinoma, endometrial carcinoma, urothelial carcinoma, squamous cell carcinoma of the head and neck, or melanoma [excluding uveal melanoma]).

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed selected solid tumor types that have progressed after treatment with standard therapies or for which there are no other appropriate therapies available.

The selected tumor types are: non-small cell lung cancer, predominantly clear cell renal cell carcinoma, endometrial carcinoma, urothelial carcinoma, squamous cell carcinoma of the head and neck, or melanoma (excluding uveal melanoma)

* At least 1 measurable target lesion according to modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Participants must have an Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) of 0 to 1.
* Adequate liver function as evidenced by bilirubin ≤1.5×ULN and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3×ULN (in the case of liver metastases ≤5×ULN). In case ALP is >3×ULN (in the absence of liver metastases) or >5×ULN (in the presence of liver metastases) AND the participant also is known to have bone metastases, the liver-specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.
* Males or females age ≥20 years at the time of informed consent
* Life expectancy of 12 weeks or more
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Prior anticancer treatment within 28 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 28 days prior to the first dose of study drugs. All toxicities related to prior treatments must be resolved to Grade ≤1 (except alopecia).
* Prior treatment with lenvatinib or any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, excluding cancer types such as melanoma and non-small cell lung cancer where prior treatment with one anti-PD-1, anti-PD-L1, or anti-PD-L2 agent is allowed
* Participants must have recovered adequately from any complications from major surgery prior to starting therapy.
* New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months
* Prolongation of QTc (Fridericia formula) interval to >480 milliseconds (ms)
* Active infection (any infection requiring systemic treatment)
* Participant is known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Known intolerance to either of the study drugs (or any of the excipients)
* History of organ allograft
* Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or has a history of interstitial lung disease
* Females who are breastfeeding or pregnant at Screening or Baseline.
* Females of childbearing potential.
* Participants must be on a stable dose of the same oral hormonal contraceptive product for at least 4 weeks before dosing with study drug and for the duration of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site 1, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitano S, Fujiwara Y, Shimizu T, Iwasa S, Yonemori K, Kondo S, Shimomura A, Koyama T, Ebata T, Ikezawa H, Hayata N, Minoshima Y, Miura T, Kubota T, Yamamoto N. A feasibility study of lenvatinib plus pembrolizumab in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2022 Dec;90(6):523-529. doi: 10.1007/s00280-022-04480-w. Epub 2022 Oct 26. PMID 36289094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 12 Jan 2017 to 15 Apr 2020.
Pre-assignment Details: A total of 11 participants were screened, of which 5 were screen failures and 6 received study treatment.
Groups:
- Lenvatinib 20 mg Plus Pembrolizumab 200 mg: Participants with selected solid tumors received oral lenvatinib at a starting dose of 20 milligram (mg), capsule, once daily in combination with intravenous pembrolizumab 200 mg every 3 weeks on a 21-day treatment cycle to confirm the dose tolerability by assessing Dose limiting toxicities (DLTs). In case of dose intolerability in Cycle 1, lenvatinib dose was reduced from 20 mg to 14 mg once daily, in combination with 200 mg pembrolizumab every 3 weeks administered up to maximum of 45 cycles or until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study (31 months).
Period: Overall Study
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Lenvatinib 20 mg Plus Pembrolizumab 200 mg: Participants with selected solid tumors received oral lenvatinib at a starting dose of 20 mg, capsule, once daily in combination with intravenous pembrolizumab 200 mg every 3 weeks on a 21-day treatment cycle to confirm the dose tolerability by assessing DLTs. In case of dose intolerability in Cycle 1, lenvatinib dose was reduced from 20 mg to 14 mg once daily, in combination with 200 mg pembrolizumab every 3 weeks administered up to maximum of 45 cycles or until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination of the study (31 months).
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerged during the time from the first dose of study drug to 30 days following the last dose of study drug, having been absent at pretreatment (Baseline) or reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. A Serious AE is any untoward medical occurrence that at any dose: resulted in death; was life threatening (that is, the participant was at immediate risk of death from the AE as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death) required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From the first dose until 30 days after the last dose (approximately 2 years 7 months)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  SAEs | 4

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: A DLT is defined as any of the following: any of the hematological or nonhematological toxicities specified in the protocol that are considered to be at least possibly related to lenvatinib and/or pembrolizumab occurring during Cycle 1; failed to administer greater than or equal to 75 percent (%) of the planned dosage of lenvatinib as a result of treatment-related toxicity during Cycle 1; participants who discontinued due to treatment-related toxicity in Cycle 1; greater than a 2-week delay in starting pembrolizumab in Cycle 2 because of a treatment-related toxicity, even if the toxicity does not meet DLT criteria.
Time Frame: Cycle 1 (Cycle length=21 days)
Population: The DLT set included all participants who completed Cycle 1 without major protocol deviation with at least 75% of study drug compliance and were assessed for DLT, and participants who experienced DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Objective Response Rate (ORR) Based on Modified Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
Description: ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) for target and non-target lesions. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in the short axis to less than 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The tumor assessment was done using number of lesions based on modified RECIST 1.1 for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or up to approximately 2 years 7 months
Population: The efficacy analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
percentage of participants | 33.3

4. Secondary Outcome: Duration of Response (DOR) Based on Modified Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
Description: DOR was defined as time from the first documented of CR or PR to the date of first documentation of disease progression (PD) (based on modified RECIST 1.1) or death (whichever occurs first). CR was defined as the disappearance of all target lesions and non-target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD for target lesion, was defined as a minimum 20% increase and a minimum 5 mm absolute increase in sum of diameters compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir was defined as lowest measure sum of diameters of target lesions at any time point from baseline onward. The tumor assessment was done using number of lesions based on modified RECIST 1.1 for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ. DOR = Date of PD/death (whichever occurs first) - Date of first CR or PR + 1.
Time Frame: as for outcome 3
Population: The efficacy analysis set included all participants who received at least 1 dose of study drug. Here overall number analyzed "N" included the participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
months | NA [16.79 to NA] — Median and upper limit of 95%CI was not estimable due to lesser number of participants with events.

5. Secondary Outcome: Cmax: Maximum Plasma Concentration of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours
Population: The PK analysis set included all participants who received at least 1 dose of lenvatinib and pembrolizumab, and had evaluable concentration data.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL) | 325 (233)

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
hours | 3.85 [1.78 to 7.02]

7. Secondary Outcome: T1/2: Terminal Half-life of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 15: 0-24 hours
Population: The PK analysis set included all participants who received at least 1 dose of lenvatinib and pembrolizumab, and had evaluable concentration data. Here overall number analyzed "N" included the participants who were evaluable for the outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
hours
  Cycle 1 Day 1 | 5.62 [5.52 to 5.71]
  Cycle 1 Day 15 | 7.26 [6.95 to 7.57]

8. Secondary Outcome: AUC(0-t): Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 3040 (1780)
  Cycle 1 Day 15 | 4280 (2600)

9. Secondary Outcome: AUC(0-inf): Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
ng*h/mL | 3880 (2090)

10. Secondary Outcome: Vz/F: Apparent Volume of Distribution at Terminal Phase of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: liter (L)
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
liter (L)
  Cycle 1 Day 1 | 41.8 (23.5)
  Cycle 1 Day 15 | 26.1 (0.636)

11. Secondary Outcome: CL/F: Apparent Total Clearance Following Oral Dosing of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours
Population: The PK analysis set included all participants who received at least 1 dose of lenvatinib and pembrolizumab, and had evaluable concentration data. Here, overall number analyzed "N" are the participants who were evaluable for the outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
liter per hour (L/hr) | 5.15 (2.78)

12. Secondary Outcome: MRT: Mean Residence Time of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
hours
  Cycle 1 Day 1 | 9.06 (0.983)
  Cycle 1 Day 15 | 11.8 (0.141)

13. Secondary Outcome: Css,Max: Maximum Observed Plasma Concentration at Steady State of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
ng/mL | 355 (319)

14. Secondary Outcome: Css,Min: Minimum Observed Plasma Concentration at Steady State of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
ng/mL | 60.1 (24.6)

15. Secondary Outcome: Tss,Max: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
hours | 7.14 [2.07 to 7.83]

16. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve Over the Dosing Interval of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 3
ng*h/mL | 6780 (1820)

17. Secondary Outcome: Clss/F: Apparent Total Clearance Following Oral Administration at Steady State of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 3
L/h | 2.95 (0.932)

18. Secondary Outcome: Css,Av: Average Steady State Plasma Concentration of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 3
ng/mL | 283 (75.8)

19. Secondary Outcome: Rac (Cmax): Accumulation Index of Cmax for Lenvatinib in Combination With Pembrolizumab
Description: Rac (Cmax) was calculated as the ratio of drug concentrations observed during a dosing interval at steady state divided by drug concentrations seen during the dosing interval after a single (first) dose. Rac (Cmax) = Css,max on Cycle 1 Day 15 / Cmax on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1: 0-24 hours and Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
ratio | 1.14 (0.376)

20. Secondary Outcome: Rac (AUC): Accumulation Index of AUC for Lenvatinib in Combination With Pembrolizumab
Description: Rac (AUC) was calculated as the ratio of drug concentrations observed during a dosing interval at steady state divided by drug concentrations seen during the dosing interval after a single (first) dose. Rac (AUC) = AUC(0-t) on Cycle 1 Day 15 / AUC(0-t) on Cycle 1 Day 1.
Time Frame: Cycle 1 Day 1: 0-24 hours and Cycle 1 Day 15: 0-24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
ratio | 1.46 (0.450)

21. Secondary Outcome: Lambda z: Terminal Phase Elimination Rate Constant of Lenvatinib in Combination With Pembrolizumab
Time Frame: Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: 1/hour
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 2
1/hour
  Cycle 1 Day 1 | 0.123 (0.00354)
  Cycle 1 Day 15 | 0.0956 (0.00573)

22. Secondary Outcome: PTF: Peak-trough Fluctuation Ratio of Lenvatinib in Combination With Pembrolizumab
Description: The peak trough fluctuation within complete dosing interval at steady state, calculated as PTF (%) = ([Cmax - Cmin]/Cav ) multiplied by 100
Time Frame: Cycle 1 Day 15: 0-24 hours
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Percentage fluctuation
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 3
Percentage fluctuation | 194 (48.8)

23. Secondary Outcome: Number of Participants Positive for Serum Anti-drug Antibodies (ADA) Status for Pembrolizumab
Time Frame: Day 1 of Cycles 1, 2, 4, 6, and 8 and every 4 cycles thereafter; within 30 days after discontinuation or until the initiation of other anticancer treatment, whichever is earlier (Cycle length=21 days); up to 31 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (approximately 2 years 7 months)
Arm/Group | Lenvatinib 20 mg Plus Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 20 mg Plus Pembrolizumab 200 mg (N=6)
Subileus (Gastrointestinal disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspergillus infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 20 mg Plus Pembrolizumab 200 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Hyperthyroidism (Endocrine disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Malaise (General disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Performance status decreased (General disorders) | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 3
Lipase increased (Investigations) | 3
Platelet count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Amylase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Electrocardiogram ST-T change (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypozincaemia (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03006887/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03006887/SAP_001.pdf